CLINICAL TRIAL: NCT00368459
Title: Raloxifene in Women With AD: Randomized Controlled Trial
Brief Title: Raloxifene for Women With Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Kaiser Permanente (Other); Indiana University (Other); Southern Illinois University (Other)
Responsible Party: Principal Investigator, Victor W. Henderson, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IA0096
Record Dates: First submitted 2006-08-22; First posted 2006-08-24 (Estimated); Results first posted 2015-04-02 (Estimated); Last update posted 2015-04-02 (Estimated); Status verified 2015-03

CONDITIONS: Alzheimer Disease
Keywords: raloxifene, women
MeSH Terms: conditions — Alzheimer Disease | interventions — Raloxifene Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- raloxifene (Experimental): oral raloxifene 120 mg once daily
  Interventions: Drug: raloxifene
- placebo (Placebo Comparator): identical appearing oral placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: raloxifene — Raloxifene is a selective estrogen receptor modulator
  Other Names: Evista
  Arms: raloxifene
Drug: Placebo — Identical appearing placebo
  Other Names: There are no other names.
  Arms: placebo

SUMMARY:
This is a multisite pilot randomized trial of raloxifene or placebo for the treatment of women with Alzheimer's disease.

DETAILED DESCRIPTION:
Raloxifene , a selective estrogen receptor modulator, has attracted attention as a potential treatment for Alzheimer's disease in women, but it has not been studied in this disorder.

To assess feasibility of large-scale efficacy trials and to obtain an initial estimate of treatment effect, study investigators plan to conduct a pilot, randomized, double blind, placebo-controlled, clinical trial of high-dose (120 mg daily) raloxifene. Eligible participants are postmenopausal women with late-onset Alzheimer's disease of mild-to-moderate severity taking a stable dose of an approved cholinesterase inhibitor. This pilot study is not designed to have power to detect significant, modest between-group differences of the magnitude provided by current FDA-approved therapies.

Study participants will be randomly allocated to oral raloxifene or identical placebo over a 12 month period. Outcomes of interest will be obtained at 6 and 12 months. The prespecified primary outcome is the change in the Alzheimer's Disease Assessment Scale, cognitive subscale (ADAS-cog), compared between groups at 12 months. Prespecified secondary outcomes include measures of global severity (Clinical Dementia Rating sum of boxes), function (Activities of Daily Living), behavior (Neuropsychiatric inventory), and other neuropsychological measures. Caregiver outcomes will be burden (Zarit burden inventory) and distress (from the Neuropsychiatric inventory).

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Post menopausal
3. Age at least 60 years
4. Eight or more years of education with a history of premorbid literacy
5. By history, fluent speaker of English
6. Dementia (DSM-IV-derived criteria) present for at least six months beginning at age 60 or older
7. Mild or moderate dementia, defined by Mini-Mental State examination (MMSE) score between 12 and 26, inclusive
8. National Institute of Neurological and Communicative Disease and the Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria for probable Alzheimer's disease (AD) based on results of a neurologist's evaluation and laboratory tests
9. Neurological history and examination within normal limits for age, except for changes consistent with AD or age
10. Modified Ischemia Scale score of 4 or less
11. Good physical health established by medical history, physical exam, and baseline laboratory tests
12. Blood pressure < 180/100 at time of entry
13. No history of, or examination evidence for, current insulin-dependent diabetes, stroke thought to impair cognition (e.g., cortical or thalamic infarct), or other focal brain lesion or neurological disorder likely to affect cognition, or other serious medical illness likely to limit participant's ability to complete study protocol
14. No history of pulmonary embolism, deep vein thrombosis, or retinal vein occlusion
15. No Diagnostic and Statistical Manual (DSM) IV criteria for Major Depressive Episode or other Axis I psychiatric disorder, other than AD, within the past year
16. Effective dose of an FDA-approved cholinesterase inhibitor for at least 6 months prior to randomization (usually donepezil 5 or 10 mg/d, rivastigmine 6 to 12 mg/d, or galantamine 16 to 24 mg/d); stable effective dose for at least 2 months prior to randomization
17. No psychotropic medication within 4 weeks of study entry or stable dose (for at least 4 weeks month) of psychotropic medications
18. No experimental mediation for the treatment of cognitive impairment associated with dementia within 2 months of study entry
19. No raloxifene within 6 months of study entry
20. No systemic estrogen, progestin, testosterone, related gonadal hormone therapy within 2 months of study entry
21. No other known contraindication to raloxifene or donepezil
22. A primary caregiver who knows the participant well and who is able to accompany her for regular assessments during the course of the study
23. Assent or consent of participant plus informed consent from participant's next of kin or legally authorized representative

Exclusion Criteria:

1. Failure to meet inclusion criteria

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2006-08; Primary Completion 2011-03 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Victor Henderson, Principal Investigator — Stanford University
Locations (4):
- United States (4):
  - Kaiser Permanente Santa Rosa, Santa Rosa, California
  - Stanford University School of Medicine, Stanford, California
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Indiana University Medical Center, Indianapolis, Indiana

RESULTS

PARTICIPANT FLOW:
Groups:
- Raloxifene: oral raloxifene 120 mg once daily
  raloxifene
Period: Overall Study
Arm/Group | Raloxifene | Placebo
Started | 21 | 21
Completed | 19 | 20
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Population: Postmenopausal women with Alzheimer's disease of mild to moderate severity
Groups:
- Total: Total of all reporting groups
Arm/Group | Raloxifene | Placebo | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 78 (4.5) | 74 (5.1) | 76 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 21 | 42
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 21 | 21 | 42
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 20 | 21 | 41
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 21 | 42

OUTCOME MEASURES:

1. Primary Outcome: Alzheimer's Disease Assessment Scale, Cognitive Subscale (ADAS-cog)
Description: ADAS-cog, change from baseline at 12 months, compared between treatment arms. The ADAS-cog is a neuropsychological battery commonly used in trials of AD patients. Error score range 0-70. For results below, positive change represents improvement/ better performance.
  For the primary outcome, as well as for secondary outcomes, the reported p-values reflect the calculated p-values.
Time Frame: 12 months
Population: Intent-to-treat
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Raloxifene | Placebo
Number analyzed (Participants) | 21 | 21
units on a scale | -3.2 (5.8) | -3.5 (8.0)
Statistical Analysis 1: Comparison: Raloxifene vs Placebo; For this pilot trial, we did not anticipate power to detect significant, clinically-meaningful between-group differences of the magnitude provided by FDA-approved AD therapies over a 12 month treatment period, but we specified that we would report trends (alpha <0.1) as a guide to future effectiveness studies; Test type: Superiority or Other; p > 0.1, ANCOVA

2. Secondary Outcome: Global Rating, Clinical Dementia Rating (CDR) Sum of Boxes
Description: Global rating of dementia severity, change from baseline at 12 months. Range 0-5. For results below, positive change represents improvement/ better performance.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Raloxifene | Placebo
Number analyzed (Participants) | 21 | 21
units on a scale | -2.6 (1.8) | -2.0 (3.2)
Statistical Analysis 1: Comparison: Raloxifene vs Placebo; Test type: Superiority or Other; p > 0.1, ANCOVA

3. Secondary Outcome: Function, Activities of Daily Living (ADL)
Description: ADL scale from the Alzheimer's Disease Cooperative Study, change from baseline at 12 months. Range 0-78. For results below, positive change represents improvement/ better performance.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Raloxifene | Placebo
Number analyzed (Participants) | 21 | 21
units on a scale | -9.1 (9.4) | -4.5 (9.5)
Statistical Analysis 1: Comparison: Raloxifene vs Placebo; Test type: Superiority or Other; p > 0.1, ANCOVA

4. Secondary Outcome: Behavior
Description: Neuropsychiatric Inventory, change from baseline at 12 months. Range 0-120. For results below, positive change represents improvement/ better performance.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Raloxifene | Placebo
Number analyzed (Participants) | 21 | 21
units on a scale | -2.3 (7.8) | -2.5 (6.3)
Statistical Analysis 1: Comparison: Raloxifene vs Placebo; Test type: Superiority or Other; p > 0.1, ANCOVA

5. Secondary Outcome: Cognitive (Neuropsychological)
Description: Global composite calculated as a weighted average of standardized scores of neuropsychological tests (weighted by the inverse intertest correlation matrix), change from baseline at 12 months. There is no theoretical maximum or minimum for this cognitive composite, with a score of 0 standardized units representing no change. For results below, positive change represents improvement/ better performance.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Raloxifene | Placebo
Number analyzed (Participants) | 21 | 21
units on a scale | -0.6 (1.8) | -1.1 (1.4)
Statistical Analysis 1: Comparison: Raloxifene vs Placebo; Test type: Superiority or Other; p > 0.1, ANCOVA

6. Secondary Outcome: ADAS-cog
Description: Change from baseline at 6 months, compared between groups. Error score range 0-70. For results below, positive change represents improvement/ better performance.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Raloxifene | Placebo
Number analyzed (Participants) | 21 | 21
units on a scale | -0.7 (4.2) | -1.8 (6.2)
Statistical Analysis 1: Comparison: Raloxifene vs Placebo; Test type: Superiority or Other; p > 0.1, ANCOVA

7. Secondary Outcome: Clinical Dementia Rating, Sum of Boxes
Description: Change from baseline at 6 months, compared between groups. Range 0-5. For results below, positive change represents improvement/ better performance.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Raloxifene | Placebo
Number analyzed (Participants) | 21 | 21
units on a scale | -0.8 (1.7) | -1.0 (2.4)
Statistical Analysis 1: Comparison: Raloxifene vs Placebo; Test type: Superiority or Other; p > 0.1, ANCOVA

8. Secondary Outcome: Function, Activities of Daily Living
Description: Change from baseline at 6 months, compared between groups. Range 0-78. For results below, positive change represents improvement/ better performance.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Raloxifene | Placebo
Number analyzed (Participants) | 21 | 21
units on a scale | -6.9 (6.7) | -0.3 (5.5)
Statistical Analysis 1: Comparison: Raloxifene vs Placebo; Test type: Superiority or Other; p < 0.01, ANCOVA — Favoring placebo, unadjusted for multiple comparisons

9. Secondary Outcome: Behavior
Description: Neuropsychiatric Inventory, change from baseline at 6 months, compared between groups. Range 0-120. For results below, positive change represents improvement/ better performance.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Raloxifene | Placebo
Number analyzed (Participants) | 21 | 21
units on a scale | -0.7 (5.6) | -2.1 (8.0)
Statistical Analysis 1: Comparison: Raloxifene vs Placebo; Test type: Superiority or Other; p > 0.1, ANCOVA

10. Secondary Outcome: Cognition (Neuropsychological)
Description: Global composite calculated as a weighted average of standardized scores of neuropsychological tests (weighted by the inverse intertest correlation matrix), change from baseline at 6 months. There is no theoretical maximum or minimum for this cognitive composite, with a score of 0 standardized units representing no change. For results below, positive change represents improvement/ better performance.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Raloxifene | Placebo
Number analyzed (Participants) | 21 | 21
units on a scale | -0.5 (1.5) | -0.6 (1.1)
Statistical Analysis 1: Comparison: Raloxifene vs Placebo; Test type: Superiority or Other; p > 0.1, ANCOVA

ADVERSE EVENTS:
Arm/Group | Raloxifene | Placebo
Serious Adverse Events (participants affected / at risk) | 2/21 | 1/21
Other Adverse Events (participants affected / at risk) | 16/21 | 13/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raloxifene (N=21) | Placebo (N=21)
colon cancer (Gastrointestinal disorders) | 1 (1) | 0 (0) — Colectomy for colon cancer diagnosed a week after study completion
agitation (Nervous system disorders) | 0 (0) | 1 (1) — Hospitalization for hallucinations and agitation
death (Nervous system disorders) | 1 (1) | 0 (0) — Ischemic stroke followed by death
hallucinations (Nervous system disorders) | 0 (0) | 1 (1) — Hospitalization for hallucinations and agitation
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Pneumonia accompanied by congestive heart failure
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raloxifene (N=21) | Placebo (N=21)
urinary tract infection (Renal and urinary disorders) | 3 (5) | 1 (1)
cold symptoms (General disorders) | 3 (3) | 2 (2)
decreased appetite (General disorders) | 3 (3) | 0 (0)
back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
arm or shoulder pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
diarrhea (Gastrointestinal disorders) | 2 (2) | 3 (3)
nausea (Gastrointestinal disorders) | 2 (2) | 2 (2)
abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
sinusitis (General disorders) | 1 (3) | 2 (4)
hallucinations (Psychiatric disorders) | 0 (0) | 3 (3)
anxiety (Psychiatric disorders) | 0 (0) | 2 (2)
paranoia (Psychiatric disorders) | 0 (0) | 3 (3)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
agitation (Psychiatric disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No